CLINICAL TRIAL: NCT00997711
Title: Evaluation of Diabetic Effects on Clinical Outcomes After Sirolimus-Eluting Stents in the AsIAN Population
Acronym: DESSIAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: Johnson & Johnson (Industry); CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0119
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
Keywords: Diabetes; death; MI; TVR
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cypher (Experimental): Sirolimus-eluting stent
  Interventions: Device: Cypher

INTERVENTIONS:
Device: Cypher — Sirolimus-eluting stents
  Other Names: Sirolimus-eluting stents

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the CYPHER SELECT™+ Sirolimus-eluting Stent (SES) in Asian diabetic patients.

DETAILED DESCRIPTION:
Study design This is a multi center, prospective, post market surveillance study of diabetic patients who underwent CYPHER SELECT™+ Sirolimus-eluting Coronary Stent implantation. For comparison, non-diabetic patients treated with SES in the concurrent period will be simultaneously enrolled.

Data will be collected in consecutive subjects treated with commercially available product and following standard clinical practice. This registry will be limited to subjects who have received only the CYPHER SELECT™+ Sirolimus-eluting Coronary Stent during the index procedure. All subjects should be treated according to the Instructions For Use (IFU) including conduct of the stenting procedure and administration of anti-platelet and diabetic medications; any other medical therapy should be provided according to local standard care. Brief study design is as depicted in the following figure.

STUDY POPULATION The registry will be conducted at approximately 15 centers in Korea where CYPHER SELECT™+ Sirolimus-eluting Coronary Stent is approved for commercial use. Data will be collected on approximately 3,600 subjects treated with the CYPHER SELECT™+ Sirolimus-eluting Coronary Stent only. Assuming the proportion of diabetic patients as 30%, approximately 1,100 diabetic patients will be enrolled. Enrolled diabetic patients are confirmed and diagnosed with Diabetes before or during the index procedure hospitalization, i.e., those receiving active treatment with an oral hypoglycemic agent or insulin, patients with diagnosis of diabetes who were on dietary therapy alone or patients with an abnormal blood glucose level after an overnight fast. Enrolled non-diabetic patients should be treated with CYPHER SELECT™+ Sirolimus-eluting Coronary Stent only.

STUDY PROCEDURE As regulated by data protection and privacy laws and in accordance with local Ethics Committee requirements, subjects will be informed and requested to grant their approval to review their medical records and collect and analyze personal medical information, while maintaining the confidentiality of the records at all times. They will be also asked to agree to be contacted during a 1-year follow-up period. Subjects will be followed at 1, 6 and 12 months, by phone call, office visit, or by contacts with primary physicians or referring cardiologists, according to each investigator's preference. Angiographic follow up will be performed at the physician's discretion. In diabetic patients, fasting glucose level and HbA1c level assessment will be performed at the index procedure and at the 12-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving CYPHER SELECT™+ Sirolimus-eluting Coronary Stent
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Any contraindication to any of the following medications: aspirin, heparin, clopidogrel, stainless steel, contrast agents, or sirolimus
* An elective surgical procedure is planned that would necessitate interruption of antiplatelet drugs during the first 6 months post enrollment.
* Cardiogenic shock
* Terminal illness with life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 953 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The composite of death, nonfatal myocardial infarction (MI), or Target- Vessel Revascularization (TVR) at 12 months post procedure. | 12-month

SECONDARY OUTCOMES:
All Death | 12-month
Cardiac death | 12 months
MI (myocardial infarction) | 12 months
Composite of death or MI | 12 months
Composite of cardiac death or MI | 12 months
Target- Vessel Revascularization (TVR) | 12 months
Target-lesion revascularization (TLR) | 12 months
Stent thrombosis (ARC criteria) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (14):
- South Korea (14):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Busan Saint Mary's Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - NHIC Ilsan Hospital, Ilsan
  - Gyeongsang Uniservity Hospital, Jinju
  - Hallym University Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea University Hospital, Seoul
  - St.Mary's Catholic Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan